CLINICAL TRIAL: NCT02852694
Title: Risk-stratified Randomized Controlled Trial in Paediatric Crohn Disease:Methotrexate Vs Azathioprine or Adalimumab for Maintaining Remission in Patients At Low or High Risk for Aggressive Disease Course, Respectively-a Treatment Strategy
Brief Title: Reduce Risk for Crohn's Disease Patients
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PIBD-Net (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01
Record Dates: First submitted 2016-06-09; First posted 2016-08-02 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Methotrexate; Adalimumab; Azathioprine; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High Risk Group (Active Comparator): subcutaneous methotrexate versus subcutaneous adalimumab
  Interventions: Drug: Methotrexate; Drug: Adalimumab
- Low risk group (Active Comparator): subcutaneous methotrexate versus oral dose of azathioprine / 6 mercaptopurine
  Interventions: Drug: Methotrexate; Drug: Azathioprine / 6 Mercaptopurine
- Ancillary (Other): the ancillary study is planned to analyse of Adalimumab treated patients from inclusion (TOP-Down) versus patients switched to Adalimumab due to failure of immunomodulator therapy (STEP-Up).
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Methotrexate — Subcutaneous methotrexate once weekly 15mg/m2 body surface area (19, 30), with a maximal dose of 25mg/week. Odansetron (Zofran) premedication (4-8mg 1Hour prior to injection) is recommended, folate acid substitution (15mg po, 3 days after Methotrexate injection, for children <20kg: 1x 5mg) is recommended.
  Arms: High Risk Group; Low risk group
Drug: Adalimumab — Subcutaneous Adalimumab started at a dose of 160mg followed by 80mg 2 weeks later and then 40mg every 2 weeks in patients over 40kg. In patients < 40kg sc doses of Adalimumab are as follows: induction 160mg/1,73m2 BSA (max 160mg), followed by 80mg/1,73m2 Body surface area (max 80mg) 2 weeks later and maintenance of 40mg/1,73m2 Body surface area (max 40mg) every 2 weeks, all doses rounded up to the nearest 5 multiplications.
  Other Names: humira
  Arms: Ancillary; High Risk Group
Drug: Azathioprine / 6 Mercaptopurine — Oral Azathioprine /6mercaptopurine at a dose of 2.5 mg/kg once daily rounded to the nearest multiplication of 12.5mg or oral 6mercaptopurine at a dose of 1.5mg/kg once daily rounded to the nearest multiplication of 12.5mg.
  Other Names: imurel / purinethol
  Arms: Low risk group

SUMMARY:
The purpose of this study is to compare the effectiveness of weekly subcutaneously administered Methotrexate for maintaining relapse-free sustained steroid/Enteral Nutrition -free 1-year remission compared with:

* daily oral Azathioprine / 6 mercaptopurine in low risk paediatric Crohn's disease
* subcutaneously administered adalimumab in high risk paediatric Crohn's disease

DETAILED DESCRIPTION:
In this randomized controlled trial PIBDNet (pediatric inflammatory bowel diseases network) aims to compare the following treatment strategy by dividing patients into two risk groups for aggressive disease evolution: the effectiveness of Methotrexate versus Azathioprine / 6 mercaptopurine for the maintenance of remission in Crohn's disease in children who are at low risk for aggressive disease and the effectiveness of Methotrexate versus adalimumab in the high risk group. PIBDNet hypothesizes that Methotrexate is superior to Azathioprine / 6 mercaptopurine for maintaining remission in Crohn's disease in the low risk strata and adalimumab is superior to Methotrexate in the high risk strata. In addition, the ancillary study is planned to analyse of Adalimumab treated patients from inclusion (TOP-Down) versus patients switched to Adalimumab due to failure of immunomodulator therapy (STEP-Up).

ELIGIBILITY:
Inclusion Criteria:

1. Children 6-17, with a new-onset Crohn Disease diagnosed using established criteria (37, 38), requiring a steroid-based or Enteral nutrition based induction therapy
2. At initial diagnosis, wPCDAI >40 or CRP>2 times upper limit at diagnosis
3. all wPCDAI scores (0-120) are possible at inclusion (patients in remission and patients with active disease)
4. Luminal active Crohn Disease (B1) with or without B2 and/or B3 disease behavior
5. Initial exposure to 5-ASA and derivate is tolerated
6. Exposure to antibiotics is tolerated
7. If one of the following criteria is present, patients are allocated to the high risk group prior randomization:

   * Complex fistulizing perianal disease
   * Panenteric disease phenotype (defined as L3 with L4b per Paris classification or L3 with deep ulcers in duodenum, stomach or oesophagus (not HP (helicobacter pylori)- or NSAID-related))
   * Severe growth impairment (height z-score <-2 or crossing 2 percentiles or more) likely related to CD
   * Significant hypoalbuminemia (<30g/l), elevated C reactive protein (CRP) (at least 2 times above normal range), or wPCDAI >12.5 despite 3 weeks of optimized induction therapy with steroids or Exclusive enteral nutrition
   * B2, B3 or B2B3 disease behavior
   * Overall cumulative disease extend of ≥60 cm
8. Informed and signed consent

Exclusion Criteria:

1. Patients with wPCDAI<42,5 at initial diagnosis, except if CRP>2 times upper limit
2. No induction therapy with steroids or enteral nutrition
3. Previous therapy with any IBD (inflammatory bowel desease) -related medications other than induction therapy as detailed in this protocol (except 5-ASA).
4. Pregnancy or refusal to use contraceptives during the study period in pubertal patients (both boys and girls) unless absolute abstinence (no sexual activity) is confirmed at each study visit. Positive pregnancy testing throughout the study will trigger prompt withdrawal of the patient from the study.
5. Lactating mothers
6. Children with perianal fistulising disease who require surgical therapy (drainage, seton placement)
7. Patients homozygous for Thiopurine methyl transferase or those with Thiopurine methyl transferase activity <6 nmol/h/ml erythrocytes or <9nmol 6MTG (6 methylthioguanine/g Hb/h), unless they qualify as high risk patients
8. Evidence of un-drained and un-controlled abscess/phlegmon
9. Contraindication to any drugs used in the trial (including intolerance/hypersensitivity or allergy to either study drug (thiopurines, methotrexate or adalimumab))
10. Current or previous malignancy
11. Serious comorbidities (such as renal insufficiency, hepatitis, respiratory insufficiency) interfering with drug therapy or interpretation of outcome parameters or will make it unlikely that the patients will finish the trial.
12. Infection with mycobacterium tuberculosis
13. Moderate to severe heart failure (NYHA classe III/IV)
14. Oral anticoagulant therapy, anti-malaria therapy
15. Live vaccines exposure (including yellow fever) less than 3 weeks prior inclusion

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Rate of sustained steroid/EEN-free remission at Month 12 | Month 12
  Rate of sustained steroid/EEN-free remission at Month 12, where sustained remission is defined as wPCDAI (weighted pediatric crohn disease activity index) ≤12.5 and CRP ≤1,5 fold the normal upper limit without a relapse since week 12.

SECONDARY OUTCOMES:
Time to first relapse | Month 12
  the goal is to compare the time of the first relapse
Remission at 12 weeks (measured by wPCDAI</=12.5 and normal CRP and being off steroids/exclusive enteral nutrition) | 12 weeks
  the goal is to compare the remission at 12 weeks
Linear height velocity | 12 months
  the goal is to compare linear height velocity
Steroid sparing effect of the regimens | 12 months
  the goal is to compare steroid sparing effect of the regimen
Comparison of toxicity of the different protocol drugs | 12 months
  Toxicity of the different protocol drugs will be compared using incidence of Adverse Events (AE) and Serious Adverse Events (SAE).
Questionnaire : health-related life of quality (IMPACT 3) between the different treatment arms | 12 months
  Health-related life of quality willl be compared between the different treatment arms, based on the IMPACT-III questionnaire, a questionnaire developed for use in pediatric inflammatory bowel disease
Clinical predictors for response, including genomic and serological markers | 12 months
  Clinical predictors for response to Study treatment will be determined, using genomic and serological markers, such as ASCA.
Predictive value of fecal calprotectin levels, CRP and other serum tests | 12 months
  the goal is to evaluate predictive value of fecal calprotectin levels, CRP and other serum tests
Questionnaire : TUMMY-CD (patient reported outcome) at month 12 | 12 months
  the goal is to evaluate questionnaire : TUMMY-CD (patient reported outcome) for all patients patients at month 12
Questionnaire : WPAI:CD Caregiver (patient reported outcome) at month 12 | 12 months
  the goal is to evauate WPAI:CD Caregiver (patient reported outcome) for all patients at month 12
Questionnaire : School Attendance (patient reported outcome) at month 12 | 12 months
  the goal is to evauate School Attendance questionnaire (patient reported outcome) for all patients at month 12
DNA pharmacogenetics (multiplex genotyping of polymorphism in drug metabolism) in relation to toxicity and response to therapy | 12 months
  the goal is to evaluate DNA pharmacogenetics (multiplex genotyping of polymorphism in drug metabolism) in relation to toxicity and response to therapy
Concentration of protocol drug (ADA or MTX) monitoring in relation to adherence, toxicity and response | 12 months
  the goal is to evaluate concentration of protocol drug (ADA or MTX) monitoring in relation to adherence, toxicity and response
6 Mercaptopurine and azathioprine metabolites monitoring : concentration of metabolites in relation to adherence, toxicity and response | 12 months
  the goal is to evaluate 6 Mercaptopurine and azathioprine metabolites monitoring : concentration of metabolites in relation to adherence, toxicity and response
Anti-adalimumab antibodies monitoring : concentration of anti-adalimumab antibodies in relation to adherence, toxicity and response | 12 months
  the goal is to evaluate anti-adalimumab antibodies monitoring : concentration of anti-adalimumab antibodies in relation to adherence, toxicity and response

CONTACTS AND LOCATIONS:
Overall Officials: Frank RUEMMELE, PhD / MD, Study Director — PIBD-Net
Locations (1):
- Hôpital Necker -Enfants Malades (Service de gastro-enterologie), Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearson DC, May GR, Fick G, Sutherland LR. Azathioprine for maintaining remission of Crohn's disease. Cochrane Database Syst Rev. 2000;(2):CD000067. doi: 10.1002/14651858.CD000067. PMID 10796482
- [Background] Faubion WA Jr, Bousvaros A. Medical therapy for refractory pediatric Crohn's disease. Clin Gastroenterol Hepatol. 2006 Oct;4(10):1199-213. doi: 10.1016/j.cgh.2006.05.031. Epub 2006 Jul 26. PMID 16872913
- [Background] Candy S, Wright J, Gerber M, Adams G, Gerig M, Goodman R. A controlled double blind study of azathioprine in the management of Crohn's disease. Gut. 1995 Nov;37(5):674-8. doi: 10.1136/gut.37.5.674. PMID 8549944
- [Background] Markowitz J, Grancher K, Kohn N, Lesser M, Daum F. A multicenter trial of 6-mercaptopurine and prednisone in children with newly diagnosed Crohn's disease. Gastroenterology. 2000 Oct;119(4):895-902. doi: 10.1053/gast.2000.18144. PMID 11040176
- [Background] D'Haens G, Geboes K, Rutgeerts P. Endoscopic and histologic healing of Crohn's (ileo-) colitis with azathioprine. Gastrointest Endosc. 1999 Nov;50(5):667-71. doi: 10.1016/s0016-5107(99)80017-0. PMID 10536324
- [Background] Chatu S, Subramanian V, Saxena S, Pollok RC. The role of thiopurines in reducing the need for surgical resection in Crohn's disease: a systematic review and meta-analysis. Am J Gastroenterol. 2014 Jan;109(1):23-34; quiz 35. doi: 10.1038/ajg.2013.402. Epub 2013 Dec 10. PMID 24322839
- [Background] Panes J, Lopez-Sanroman A, Bermejo F, Garcia-Sanchez V, Esteve M, Torres Y, Domenech E, Piqueras M, Gomez-Garcia M, Gutierrez A, Taxonera C, Sans M; AZTEC Study Group. Early azathioprine therapy is no more effective than placebo for newly diagnosed Crohn's disease. Gastroenterology. 2013 Oct;145(4):766-74.e1. doi: 10.1053/j.gastro.2013.06.009. Epub 2013 Jun 13. PMID 23770132
- [Background] Cosnes J, Bourrier A, Laharie D, Nahon S, Bouhnik Y, Carbonnel F, Allez M, Dupas JL, Reimund JM, Savoye G, Jouet P, Moreau J, Mary JY, Colombel JF; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif (GETAID). Early administration of azathioprine vs conventional management of Crohn's Disease: a randomized controlled trial. Gastroenterology. 2013 Oct;145(4):758-65.e2; quiz e14-5. doi: 10.1053/j.gastro.2013.04.048. Epub 2013 Apr 30. PMID 23644079
- [Background] Alfadhli AA, McDonald JW, Feagan BG. Methotrexate for induction of remission in refractory Crohn's disease. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD003459. doi: 10.1002/14651858.CD003459.pub2. PMID 15674908
- [Background] Feagan BG, Fedorak RN, Irvine EJ, Wild G, Sutherland L, Steinhart AH, Greenberg GR, Koval J, Wong CJ, Hopkins M, Hanauer SB, McDonald JW. A comparison of methotrexate with placebo for the maintenance of remission in Crohn's disease. North American Crohn's Study Group Investigators. N Engl J Med. 2000 Jun 1;342(22):1627-32. doi: 10.1056/NEJM200006013422202. PMID 10833208
- [Background] Feagan BG, Rochon J, Fedorak RN, Irvine EJ, Wild G, Sutherland L, Steinhart AH, Greenberg GR, Gillies R, Hopkins M, et al. Methotrexate for the treatment of Crohn's disease. The North American Crohn's Study Group Investigators. N Engl J Med. 1995 Feb 2;332(5):292-7. doi: 10.1056/NEJM199502023320503. PMID 7816064
- [Background] Kozarek RA, Patterson DJ, Gelfand MD, Botoman VA, Ball TJ, Wilske KR. Methotrexate induces clinical and histologic remission in patients with refractory inflammatory bowel disease. Ann Intern Med. 1989 Mar 1;110(5):353-6. doi: 10.7326/0003-4819-110-5-353. PMID 2492786
- [Background] Holtmann MH, Krummenauer F, Claas C, Kremeyer K, Lorenz D, Rainer O, Vogel I, Bocker U, Bohm S, Buning C, Duchmann R, Gerken G, Herfarth H, Lugering N, Kruis W, Reinshagen M, Schmidt J, Stallmach A, Stein J, Sturm A, Galle PR, Hommes DW, D'Haens G, Rutgeerts P, Neurath MF. Long-term effectiveness of azathioprine in IBD beyond 4 years: a European multicenter study in 1176 patients. Dig Dis Sci. 2006 Sep;51(9):1516-24. doi: 10.1007/s10620-005-9037-5. Epub 2006 Aug 22. PMID 16927148
- [Background] Lemann M, Mary JY, Colombel JF, Duclos B, Soule JC, Lerebours E, Modigliani R, Bouhnik Y; Groupe D'Etude Therapeutique des Affections Inflammatoires du Tube Digestif. A randomized, double-blind, controlled withdrawal trial in Crohn's disease patients in long-term remission on azathioprine. Gastroenterology. 2005 Jun;128(7):1812-8. doi: 10.1053/j.gastro.2005.03.031. PMID 15940616
- [Background] Lemann M, Zenjari T, Bouhnik Y, Cosnes J, Mesnard B, Rambaud JC, Modigliani R, Cortot A, Colombel JF. Methotrexate in Crohn's disease: long-term efficacy and toxicity. Am J Gastroenterol. 2000 Jul;95(7):1730-4. doi: 10.1111/j.1572-0241.2000.02190.x. PMID 10925976
- [Background] Ardizzone S, Bollani S, Manzionna G, Imbesi V, Colombo E, Bianchi Porro G. Comparison between methotrexate and azathioprine in the treatment of chronic active Crohn's disease: a randomised, investigator-blind study. Dig Liver Dis. 2003 Sep;35(9):619-27. doi: 10.1016/s1590-8658(03)00372-4. PMID 14563183
- [Background] Oren R, Moshkowitz M, Odes S, Becker S, Keter D, Pomeranz I, Shirin H, Reisfeld I, Broide E, Lavy A, Fich A, Eliakim R, Patz J, Villa Y, Arber N, Gilat T. Methotrexate in chronic active Crohn's disease: a double-blind, randomized, Israeli multicenter trial. Am J Gastroenterol. 1997 Dec;92(12):2203-9. PMID 9399753
- [Background] Ravikumara M, Hinsberger A, Spray CH. Role of methotrexate in the management of Crohn disease. J Pediatr Gastroenterol Nutr. 2007 Apr;44(4):427-30. doi: 10.1097/MPG.0b013e3180320689. PMID 17414138
- [Background] Mack DR, Young R, Kaufman SS, Ramey L, Vanderhoof JA. Methotrexate in patients with Crohn's disease after 6-mercaptopurine. J Pediatr. 1998 May;132(5):830-5. doi: 10.1016/s0022-3476(98)70313-0. PMID 9602195
- [Background] Uhlen S, Belbouab R, Narebski K, Goulet O, Schmitz J, Cezard JP, Turck D, Ruemmele FM. Efficacy of methotrexate in pediatric Crohn's disease: a French multicenter study. Inflamm Bowel Dis. 2006 Nov;12(11):1053-7. doi: 10.1097/01.mib.0000235103.47280.bb. PMID 17075346
- [Background] Turner D, Grossman AB, Rosh J, Kugathasan S, Gilman AR, Baldassano R, Griffiths AM. Methotrexate following unsuccessful thiopurine therapy in pediatric Crohn's disease. Am J Gastroenterol. 2007 Dec;102(12):2804-12; quiz 2803, 2813. doi: 10.1111/j.1572-0241.2007.01474.x. PMID 18042110
- [Background] Hyams J, Crandall W, Kugathasan S, Griffiths A, Olson A, Johanns J, Liu G, Travers S, Heuschkel R, Markowitz J, Cohen S, Winter H, Veereman-Wauters G, Ferry G, Baldassano R; REACH Study Group. Induction and maintenance infliximab therapy for the treatment of moderate-to-severe Crohn's disease in children. Gastroenterology. 2007 Mar;132(3):863-73; quiz 1165-6. doi: 10.1053/j.gastro.2006.12.003. Epub 2006 Dec 3. PMID 17324398
- [Background] Hyams JS, Griffiths A, Markowitz J, Baldassano RN, Faubion WA Jr, Colletti RB, Dubinsky M, Kierkus J, Rosh J, Wang Y, Huang B, Bittle B, Marshall M, Lazar A. Safety and efficacy of adalimumab for moderate to severe Crohn's disease in children. Gastroenterology. 2012 Aug;143(2):365-74.e2. doi: 10.1053/j.gastro.2012.04.046. Epub 2012 May 2. PMID 22562021
- [Background] D'Haens G, Baert F, van Assche G, Caenepeel P, Vergauwe P, Tuynman H, De Vos M, van Deventer S, Stitt L, Donner A, Vermeire S, Van De Mierop FJ, Coche JR, van der Woude J, Ochsenkuhn T, van Bodegraven AA, Van Hootegem PP, Lambrecht GL, Mana F, Rutgeerts P, Feagan BG, Hommes D; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Early combined immunosuppression or conventional management in patients with newly diagnosed Crohn's disease: an open randomised trial. Lancet. 2008 Feb 23;371(9613):660-667. doi: 10.1016/S0140-6736(08)60304-9. PMID 18295023
- [Background] Prideaux L, De Cruz P, Ng SC, Kamm MA. Serological antibodies in inflammatory bowel disease: a systematic review. Inflamm Bowel Dis. 2012 Jul;18(7):1340-55. doi: 10.1002/ibd.21903. Epub 2011 Nov 8. PMID 22069240
- [Background] North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition; Colitis Foundation of America; Bousvaros A, Antonioli DA, Colletti RB, Dubinsky MC, Glickman JN, Gold BD, Griffiths AM, Jevon GP, Higuchi LM, Hyams JS, Kirschner BS, Kugathasan S, Baldassano RN, Russo PA. Differentiating ulcerative colitis from Crohn disease in children and young adults: report of a working group of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition and the Crohn's and Colitis Foundation of America. J Pediatr Gastroenterol Nutr. 2007 May;44(5):653-74. doi: 10.1097/MPG.0b013e31805563f3. PMID 17460505
- [Background] Winther KV, Fogh P, Thomsen OO, Brynskov J. Inflammatory bowel disease (ulcerative colitis and Crohn's disease): diagnostic criteria and differential diagnosis. Drugs Today (Barc). 1998 Nov;34(11):935-42. doi: 10.1358/dot.1998.34.11.487477. PMID 14743262
- [Background] Rosh JR. Methotrexate. In: Mamula P, Baldassano RN, Markowitz JE, editors. Pediatric inflammatory bowel disease2007. p. In press.
- [Background] Ruemmele FM, Veres G, Kolho KL, Griffiths A, Levine A, Escher JC, Amil Dias J, Barabino A, Braegger CP, Bronsky J, Buderus S, Martin-de-Carpi J, De Ridder L, Fagerberg UL, Hugot JP, Kierkus J, Kolacek S, Koletzko S, Lionetti P, Miele E, Navas Lopez VM, Paerregaard A, Russell RK, Serban DE, Shaoul R, Van Rheenen P, Veereman G, Weiss B, Wilson D, Dignass A, Eliakim A, Winter H, Turner D; European Crohn's and Colitis Organisation; European Society of Pediatric Gastroenterology, Hepatology and Nutrition. Consensus guidelines of ECCO/ESPGHAN on the medical management of pediatric Crohn's disease. J Crohns Colitis. 2014 Oct;8(10):1179-207. doi: 10.1016/j.crohns.2014.04.005. Epub 2014 Jun 6. PMID 24909831
- [Background] Froslie KF, Jahnsen J, Moum BA, Vatn MH; IBSEN Group. Mucosal healing in inflammatory bowel disease: results from a Norwegian population-based cohort. Gastroenterology. 2007 Aug;133(2):412-22. doi: 10.1053/j.gastro.2007.05.051. Epub 2007 Jun 2. PMID 17681162
- [Background] Vernier-Massouille G, Balde M, Salleron J, Turck D, Dupas JL, Mouterde O, Merle V, Salomez JL, Branche J, Marti R, Lerebours E, Cortot A, Gower-Rousseau C, Colombel JF. Natural history of pediatric Crohn's disease: a population-based cohort study. Gastroenterology. 2008 Oct;135(4):1106-13. doi: 10.1053/j.gastro.2008.06.079. Epub 2008 Jul 3. PMID 18692056
- [Background] Van Limbergen J, Russell RK, Drummond HE, Aldhous MC, Round NK, Nimmo ER, Smith L, Gillett PM, McGrogan P, Weaver LT, Bisset WM, Mahdi G, Arnott ID, Satsangi J, Wilson DC. Definition of phenotypic characteristics of childhood-onset inflammatory bowel disease. Gastroenterology. 2008 Oct;135(4):1114-22. doi: 10.1053/j.gastro.2008.06.081. Epub 2008 Jul 3. PMID 18725221
- [Background] Pigneur B, Escher J, Elawad M, Lima R, Buderus S, Kierkus J, Guariso G, Canioni D, Lambot K, Talbotec C, Shah N, Begue B, Rieux-Laucat F, Goulet O, Cerf-Bensussan N, Neven B, Ruemmele FM. Phenotypic characterization of very early-onset IBD due to mutations in the IL10, IL10 receptor alpha or beta gene: a survey of the Genius Working Group. Inflamm Bowel Dis. 2013 Dec;19(13):2820-8. doi: 10.1097/01.MIB.0000435439.22484.d3. PMID 24216686
- [Background] Pigneur B, Seksik P, Viola S, Viala J, Beaugerie L, Girardet JP, Ruemmele FM, Cosnes J. Natural history of Crohn's disease: comparison between childhood- and adult-onset disease. Inflamm Bowel Dis. 2010 Jun;16(6):953-61. doi: 10.1002/ibd.21152. PMID 19834970
- [Background] Ruemmele FM, Lachaux A, Cezard JP, Morali A, Maurage C, Ginies JL, Viola S, Goulet O, Lamireau T, Scaillon M, Breton A, Sarles J; Groupe Francophone d'Hepatologie, Gastroenterologie et Nutrition Pediatrique. Efficacy of infliximab in pediatric Crohn's disease: a randomized multicenter open-label trial comparing scheduled to on demand maintenance therapy. Inflamm Bowel Dis. 2009 Mar;15(3):388-94. doi: 10.1002/ibd.20788. PMID 19023899
- [Background] Sharma S, Eckert D, Hyams JS, Mensing S, Thakkar RB, Robinson AM, Rosh JR, Ruemmele FM, Awni WM. Pharmacokinetics and exposure-efficacy relationship of adalimumab in pediatric patients with moderate to severe Crohn's disease: results from a randomized, multicenter, phase-3 study. Inflamm Bowel Dis. 2015 Apr;21(4):783-92. doi: 10.1097/MIB.0000000000000327. PMID 25723614
- [Background] Khanna R, Bressler B, Levesque BG, Zou G, Stitt LW, Greenberg GR, Panaccione R, Bitton A, Pare P, Vermeire S, D'Haens G, MacIntosh D, Sandborn WJ, Donner A, Vandervoort MK, Morris JC, Feagan BG; REACT Study Investigators. Early combined immunosuppression for the management of Crohn's disease (REACT): a cluster randomised controlled trial. Lancet. 2015 Nov 7;386(10006):1825-34. doi: 10.1016/S0140-6736(15)00068-9. Epub 2015 Sep 3. PMID 26342731
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Torres J, Caprioli F, Katsanos KH, Lobaton T, Micic D, Zeroncio M, Van Assche G, Lee JC, Lindsay JO, Rubin DT, Panaccione R, Colombel JF. Predicting Outcomes to Optimize Disease Management in Inflammatory Bowel Diseases. J Crohns Colitis. 2016 Dec;10(12):1385-1394. doi: 10.1093/ecco-jcc/jjw116. Epub 2016 Jun 9. PMID 27282402
- [Derived] Neyt M, Christiaens A, Aloi M, de Ridder L, Croft NM, Koletzko S, Levine A, Turner D, Russell RK, Ruemmele FM, Veereman G. Identifying Health Economic Considerations to Include in the Research Protocol of a Randomized Controlled Trial (the REDUCE-RISK Trial): Systematic Literature Review and Assessment. JMIR Form Res. 2021 Jan 25;5(1):e13888. doi: 10.2196/13888. PMID 33492239
- [Derived] Harris RE, Aloi M, de Ridder L, Croft NM, Koletzko S, Levine A, Turner D, Veereman G, Neyt M, Bigot L, Ruemmele FM, Russell RK; PIBD SETQuality consortium and PIBDnet. Protocol for a multinational risk-stratified randomised controlled trial in paediatric Crohn's disease: methotrexate versus azathioprine or adalimumab for maintaining remission in patients at low or high risk for aggressive disease course. BMJ Open. 2020 Jul 1;10(7):e034892. doi: 10.1136/bmjopen-2019-034892. PMID 32611737